CLINICAL TRIAL: NCT05645523
Title: Feasibility and Safety of Indocyanine Green (ICG) Guided Sentinel Lymph Node Mapping for Pediatric Visceral Solid Tumors
Brief Title: Indocyanine Green (ICG) Guided Sentinel Lymph Node Mapping for Pediatric Visceral Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VISCERALx; NCI-2022-10202 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: Indocyanine Green; Sentinel Lymph Node Mapping; Pediatric; Young Adult
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Indocyanine green (ICG) (Experimental): Participants will receive Indocyanine green intraoperatively.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Given in to the vein (IV)
  Other Names: IC-GREEN™; ICG

SUMMARY:
The purpose of the study is to find out the usefulness and safety of a dye called Indocyanine Green (ICG for short). This dye will be used to help the surgeon find lymph nodes draining solid tumors inside the abdomen that need to be removed. This may also help the surgeon to find if the cancer has moved to other lymph nodes outside of the known area.

Primary Objectives

* To determine the percentage of patients in whom Indocyanine Green (ICG)-guided sentinel lymph node (SLN) mapping was successful at the time of retroperitoneal lymph node dissection for staging of visceral solid tumors.
* To determine the percentage of patients with grade 3 or higher adverse events related to ICG use.

DETAILED DESCRIPTION:
During surgery, participants will be given the dye to help the doctor see the lymph nodes to be removed. Pictures or a video of the procedure will be done. The number of lymph nodes removed will be recorded. After surgery, the lymph nodes will be examined.

Participants will be followed for up to 24 hours after surgery to determine if there were any side effects from the dye.

ELIGIBILITY:
Inclusion Criteria:

* Any patient under the age of 21 years with visceral pediatric solid tumor suspected to be Wilms tumor or para-testicular rhabdomyosarcoma requiring retroperitoneal lymph node dissection.

Exclusion Criteria:

* Subjects with a history of iodide allergies.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Pregnant female.
* Patients with extensive prior surgery at the primary site or nodal basin expected to affect the lymphatic drainage.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in whom Indocyanine Green (ICG)-guided sentinel lymph node (SLN) mapping was successful | During surgery (Intraoperatively)
  The estimated percentage of ICG identification and its confidence interval (CI) based on the Pearson-Klopper method exact method will be calculated.
Percentage of patients with grade 3 or higher adverse events related to ICG use | From the time of ICG administration to 24 hours after surgery (post-surgery)
  Adverse Events will be captured from the time of ICG administration to 24 hours post-surgery. Adverse Events will be graded by this scale: the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davidoff, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Lurie Children's Hospital, Chicago, Illinois
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols